CLINICAL TRIAL: NCT02637960
Title: A Randomised, Double-blind, Placebo-controlled, Multi-centre Study to Investigate the Efficacy and Safety of Fedovapagon in the Treatment of Nocturia in Men With Benign Prostatic Hyperplasia (BPH) (EQUINOC Study)
Brief Title: Efficacy Study of Fedovapagon for Nocturia in Men With Benign Prostatic Hyperplasia (BPH)
Acronym: EQUINOC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 483-013
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Nocturia
Keywords: VA106483, fedovapagon, BPH, nocturia, EQUINOC
MeSH Terms: conditions — Nocturia; Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fedovapagon 2 mg (Experimental): One daily dose of 2 mg fedovapagon for 12 weeks
  Interventions: Drug: Fedovapagon 2 mg
- Placebo matched to fedovapagon (Experimental): One daily dose of placebo (matched to fedovapagon) for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fedovapagon 2 mg — One daily dose of 2 mg fedovapagon for 12 weeks
  Arms: Fedovapagon 2 mg
Drug: Placebo — One daily dose of placebo (matched to fedovapagon) for 12 weeks
  Arms: Placebo matched to fedovapagon

SUMMARY:
This study will investigate the efficacy and safety of fedovapagon in the treatment of nocturia in men with BPH.

DETAILED DESCRIPTION:
Fedovapagon is a selective vasopressin V2 receptor (V2R) agonist that has an antidiuretic effect through stimulation of V2 receptors in the kidney and is being developed for the treatment of nocturia. Nocturia, defined as the complaint that the individual has to wake at night one or more times to void, is a common condition and shows an age-dependent increase in both prevalence and severity (number of nocturnal voids). It has a significant detrimental impact on the quality of life in patients with benign prostatic hyperplasia (BPH).

The purpose of this study is to determine the efficacy and safety of fedovapagon in the treatment of nocturia with BPH.

ELIGIBILITY:
Inclusion Criteria:

* Adult males ≥18 years [no upper limit]
* Benign prostatic hyperplasia
* Persistent nocturia despite previous lifestyle modification advice including appropriate fluid management
* Serum sodium not below lower limit of normal prior to randomization
* Provide signed and dated informed consent before any study-specific procedures are conducted.
* Able to comply with the requirements of the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in the mean number of night-time voids | 12 weeks
Change in mean patient reported nocturia bother score | 12 weeks

SECONDARY OUTCOMES:
Change in the mean number of night-time voids | 1 week
Change in the mean number of night-time voids | 4 weeks
Change in mean patient reported nocturia bother score | 1 week
Change in mean patient reported nocturia bother score | 4 weeks
Change in mean night-time urine production, absolute and as a proportion of 24 hour urine production | 2 months
Change in mean functional bladder capacity | 2 months
Change in International Prostate Symptom Score (IPSS) | 4 weeks
Change in International Prostate Symptom Score (IPSS) | 12 weeks
Change in N-QOL Score | 4 weeks
Change in N-QOL Score | 12 weeks
Number and type of Adverse Events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gittelman, MD, FACS, Principal Investigator — South Florida Medical Research
Locations (48):
- United States (48):
  - Vantia Investigative Center, Anniston, Alabama
  - Vantia Investigative Center, Goodyear, Arizona
  - Vantia Investigative Center, Lincoln, California
  - Vantia Investigative Center, Murrieta, California
  - Vantia Investigative Center, San Diego, California
  - Vantia Investigative Center, Aventura, Florida
  - Vantia Investigative Center, Bradenton, Florida
  - Vantia Investigative Center, Clearwater, Florida
  - Vantia Investigative Center, Coral Gables, Florida
  - Vantia Investigative Center, DeLand, Florida
  - Vantia Investigative Center, Hialeah, Florida
  - Vantia Investigative Center, Miami, Florida
  - Vantia Investigative Center, Ocala, Florida
  - Vantia Investigative Center, Pembroke Pines, Florida
  - Vantia Investigative Center, St. Petersburg, Florida
  - Vantia Investigative Center, Tampa, Florida
  - Vantia Investigative Center, Avon, Indiana
  - Vantia Investigative Center, Topeka, Kansas
  - Vantia Investigative Center, Wichita, Kansas
  - Vantia Investigative Center, Greenbelt, Maryland
  - Vantia Investigative Center, Missoula, Montana
  - Vantia Investigative Center, Omaha, Nebraska
  - Vantia Investigative Center, Englewood, New Jersey
  - Vantia Investigative Center, Lawrenceville, New Jersey
  - Vantia Investigative Center, Albuquerque, New Mexico
  - Vantia Investigative Center, Garden City, New York
  - Vantia Investigative Center, New York, New York
  - Vantia Investigative Center, Newburgh, New York
  - Vantia Investigative Center, Poughkeepsie, New York
  - Vantia Investigative Center, Cary, North Carolina
  - Vantia Investigative Center, Concord, North Carolina
  - Vantia Investigative Center, High Point, North Carolina
  - Vantia Investigative Center, Raleigh, North Carolina
  - Vantia Investigative Center, Wilmington, North Carolina
  - Vantia Investigative Center, Winston-Salem, North Carolina
  - Vantia Investigative Center, Akron, Ohio
  - Vantia Investigative Center, Warwick, Rhode Island
  - Vantia Investigative Center, Charleston, South Carolina
  - Vantia Investigative Center, Greer, South Carolina
  - Vantia Investigative Center, Mt. Pleasant, South Carolina
  - Vantia Investigative Center, Bristol, Tennessee
  - Vantia Investigative Center, Dallas, Texas
  - Vantia Investigative Center, Houston, Texas
  - Vantia Investigative Center, San Antonio, Texas
  - Vantia Investigative Center, Clinton, Utah
  - Vantia Investigative Center, Ogden, Utah
  - Vantia Investigative Center, Salt Lake City, Utah
  - Vantia Investigative Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No